CLINICAL TRIAL: NCT05872503
Title: Observational Study of Rates of Prostate Cancer Diagnosis in Men of African Ancestry Using MRI and MRI Guided Biopsy
Brief Title: Study of Rates of Prostate Cancer Diagnosis in Men of African Ancestry Using MRI and MRI Guided Biopsy
Status: Terminated | Type: Observational
Why Stopped: Slow accrual.
Sponsor: National Cancer Institute (NCI) (NIH)
Responsible Party: Sponsor
Organization: National Institutes of Health Clinical Center (CC) (NIH)
Other Study IDs: 10001567; 001567-C
Record Dates: First submitted 2023-05-20; First posted 2023-05-24 (Actual); Last update posted 2025-07-10 (Actual); Status verified 2025-07

CONDITIONS: Prostate Specific Antigens; Positive Digital Rectal Examination; Strong Family History of Prostate Cancer; Prostatic Neoplasms
Keywords: Health Disparity; Multiparametric MRI; MRI-Guided Biopsy; Prostate Cancer
MeSH Terms: conditions — Prostatic Neoplasms

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (1):
- Cohort 1: Participants of African Ancestry with elevated serum prostate specific antigen of (Bullet)3ng/ml or positive digital rectal examination or strong family history.

SUMMARY:
Background:

Prostate cancer (PCa) is one of the most common cancers in American men; it is a leading cause of death. Men of African ancestry have a higher rate of prostate cancer, and a higher likelihood of death, compared to men of European ancestry. The reasons for these higher rates are not known; they may include genetic and environmental factors. Better screening methods are needed.

Objective:

To test an imaging technology called multiparametric magnetic resonance imaging (mpMRI) for detecting prostate cancer in men of African ancestry.

Eligibility:

Men of African ancestry aged 35 years or older with prostate cancer and/or a strong family history of prostate cancer.

Design:

Participants will be screened. They will have a physical exam with blood and urine tests.

Participants will have an mpMRI. They will lie on a narrow bed that slides into a large cylinder. They will lie still for about 45 minutes. They will hear loud noises during the scan; they may wear earplugs or headphones to muffle the sound. Some participants may have a dye injected into a vein.

If the scan indicates participants risk of prostate cancer is medium or high, they will have a biopsy: The area will be numbed, and samples of tissue will be removed from the prostate. The biopsy will be done within 6 months.

If the scan indicates participants risk of prostate cancer is low, they will not have a biopsy.

All participants will be followed for 5 years. They and/or their local doctors will be contacted once a year for follow-up. Additional mpMRIs may be recommended.

DETAILED DESCRIPTION:
Background:

* Prostate cancer (PCa) is the most common non-dermatologic malignancy among American men and is a leading cause of cancer mortality. Men of African Ancestry (AA) have a 1.8- fold higher incidence of prostate cancer and a 2.2-fold higher likelihood of death when compared to men of European Ancestry. The predominant factor in the increased death rate is the increased incidence of cancer. The underlying reasons for the increase in incidence are controversial but likely include genetic and environmental factors.
* One strategy to counteract the effects of increased cancer incidence in a given patient population is to utilize earlier and/or more intense screening as it leads to earlier diagnosis and potentially better outcomes.
* Multiparametric MRI (mpMRI) is a proven useful tool in the diagnosis of prostate cancer but access to high quality mpMRI in communities of color is often limited.
* For individuals who are members of communities of color, high quality prostate MRI is a limited resource and insurance coverage is often denied. Given the high risk of prostate cancer in these communities, the benefits of screening with mpMRI and mpMRI guided biopsies could be significant as it could enable earlier diagnosis.

Objective:

-To compare results of mpMRI and mpMRI guided biopsy in diagnosing clinically significant prostate cancer between men of African Ancestry from hospitals providing medical care for communities of color (e.g., Howard University Hospital, Washington Hospital Center) with the population of self-referred participants seen at NIH who are mostly of European Ancestry.

Eligibility:

* Age >35 years
* Self-identified men of African Ancestry
* Elevated serum prostate specific antigen (PSA) of >=3ng/ml and/or positive digital rectal examination and/or strong family history of cancer

Design:

* This is a prospective single arm observational study.
* Up to 345 prostate biopsy na(SqrRoot) ve participants will be recruited to evaluate the use of mpMRI and mpMRI guided biopsy in diagnosing localized clinically significant prostate cancer among men of African Ancestry.
* Study participants will be referred by hospitals that mainly provide medical care for communities of color (e.g., Howard University Hospital, Washington Hospital Center).
* Participants will undergo a state-of-the-art mpMRI of the prostate in the Molecular Imaging Branch, NCI.
* If a suitable lesion (Prostate Imaging Reporting and Data System (PI-RADS >=3) is identified, mpMRI/transrectal ultrasound (TRUS) fusion guided and standard of care systematic TRUS guided biopsies of the prostate will be performed within 6 months after the mpMRI. Participants with no PI-RADS score >=3 lesions at baseline mpMRI will not have a biopsy but will be followed for 5 years.
* Participants with a positive baseline mpMRI will be in follow-up for 5 years and have phone/virtual visits occurring annually. Prostate cancer related records and overall 5 year survival status of the participants will be monitored during these follow up visits. If clinically indicated and per referring physician, additional follow up MRIs and PSAs may be obtained annually or bi-annually.

ELIGIBILITY:
* INCLUSION CRITERIA:
* Age >35 years.
* Men self-identified as being of African Ancestry.
* Elevated serum prostate specific antigen of >=3ng/ml and/or positive digital rectal examination and/or strong family history of prostate cancer (at least 1 first or second degree male relative).
* ECOG performance status <=2.
* Ability of participant to understand and the willingness to sign a written informed consent document.
* Must be co-enrolled in protocols 16-C-0010 and/or 18-C-0017.

EXCLUSION CRITERIA:

* Prior prostate biopsy.
* Prior radiotherapy or surgery for prostate cancer.
* Prior or ongoing hormonal therapy or chemotherapy (e.g., docetaxel) for prostate cancer.
* Participants unwilling or unable to undergo MRI, including participants with contraindications to MRI.
* Participants unwilling or unable to undergo biopsy, including participants with contraindications to biopsy.

Ages: 35 Years to 120 Years | Sex: Male | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: It is expected that participants for this single site study will be enrolled through referral from primary care clinics of local hospitals serving communities of color.
Sampling Method: Non-Probability Sample
Enrollment: 3 (Actual)
Dates: Start 2024-03-20 (Actual); Primary Completion 2024-09-10 (Actual); Study Completion 2024-09-10 (Actual)

PRIMARY OUTCOMES:
Cancer detection rate | mpMRI performed at baseline visit 1 and mpMRI guided biopsy performed within 6 months after that in participants with PI-RADS score >=3.
  To compare results of mpMRI and mpMRI guided biopsy in diagnosing clinically significant prostate cancer between men of African Ancestry (AA) from hospitals providing medical care for communities of color (e.g., Howard University Hospital, Washington Hospital Center) with the population of self-referred participants seen at NIH who are mostly Caucasian.

SECONDARY OUTCOMES:
Provide a summary of the report to local health insurance companies | End of study
  To provide data to insurers that supports reimbursement of MRI in men of African Ancestry in order to improve access to care.
Sensitivity and Area under the curve (AUC) | Study duration
  To use and further develop artificial intelligence (AI) algorithms to predict for clinically significant prostate cancer in men of African Ancestry based on MRI and clinical features as well as genomic risk scores.
Prostate cancer status and overall survival in mid-term (5 years) follow up | 5 years
  To evaluate prostate cancer status and overall survival in mid-term (5 years) follow up course after baseline MRI
Genomic sequencing findings | Baseline visit 1 and visit 2.
  To evaluate genomic sequencing of diagnosed tumors in men of African Ancestry and compare it to the population of self-referred participants to the NCI which is predominantly Caucasian.
Polygenic risk score | Study duration
  To evaluate the predictive value of the polygenic risk score (PRS) in predicting clinically significant prostate cancer in men of African Ancestry.

CONTACTS AND LOCATIONS:
Overall Officials: Ismail B Turkbey, M.D., Principal Investigator — National Cancer Institute (NCI)
Locations (1):
- National Institutes of Health Clinical Center, Bethesda, Maryland, United States

IPD SHARING:
Plan to Share IPD: Yes
All IPD recorded in the medical record will be shared with intramural investigators upon request. In addition, all large scale genomic sequencing data will be shared with subscribers to dbGaP.
Supporting Information: Study Protocol, SAP, ICF
Time Frame: Clinical data available during the study and indefinitely. Genomic data are available once genomic data are uploaded per protocol GDS plan for as long as database is active.
Access Criteria: Clinical data will be made available via subscription to BTRIS and with the permission of the study PI. Genomic data are made available via dbGaP through requests to the data custodians.

REFERENCES:
- See also: NIH Clinical Center Detailed Web Page — https://clinicalstudies.info.nih.gov/cgi/detail.cgi?B_001567-C.html